CLINICAL TRIAL: NCT05983900
Title: Clinical Evaluation and Antimicrobial Effect of Papain Based Chemo-mechanical Caries Removal Agents in Young Permanent Molars (A Randomized Controlled Clinical Trial)
Brief Title: Clinical Evaluation and Antimicrobial Effect of Papain Based Chemo-mechanical Caries Removal Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9197358
Record Dates: First submitted 2023-06-09; First posted 2023-08-09 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Papacarie

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BRIX 3000 (Experimental): brix 3000 used
  Interventions: Procedure: BRIX3000
- Papacarie (Active Comparator): papacarie duo used
  Interventions: Procedure: papacarie
- Hand excavation (Active Comparator): hand excavation used
  Interventions: Procedure: hand excavation

INTERVENTIONS:
Procedure: BRIX3000 — chemo-mechanical caries removal agent
  Arms: BRIX 3000
Procedure: papacarie — chemo-mechanical caries removal agent
  Arms: Papacarie
Procedure: hand excavation — mechanical caries removal
  Arms: Hand excavation

SUMMARY:
Minimally invasive dentistry continues to gain importance, especially in the treatment of permanent teeth with deep caries lesions and immature roots. Chemo-mechanical caries removal (CMCR) is an alternative to the conventional method and consists of the application of a proteolytic substance that softens carious dentin tissue and facilitates its removal using manual instruments. This method can be employed without the use of local anesthesia or burs, thereby preserving sound dental tissue.

The trial aim to assess the clinical performance of Brix 3ooo and Papacarie duo gel as chemo-mechanical caries removal agents (CMCR), their performance in terms of time required for the caries removal, patient subjective pain reaction, their radiographic success and their antimicrobial effect in comparison with Atraumatic Restorative Treatment (ART) hand excavation method for caries removal.

The trial will include 108 children with age ranging between 8 and 10 years old who have at least one carious first permanent molar will be randomly divided into three groups. A three-arm randomized clinical trial where test groups, group I, caries removal will be using Brix 3000, and group II Papacarie duo will be used, while the control group hand excavation will be the method of caries removal. Dentin samples of three groups will be taken prior to and following caries removal. The total viable streptococci and lactobacilli count will be determined and expressed as colony forming units per milliliter (CFU). The time required for caries removal with each method will be calculated and the subjective pain reaction following each method will be recorded. After complete caries removal step, it will be followed by restoration with glass ionomer restoration. Patients will be followed up at 3-, 6- and 12-month intervals to determine the clinical success and at 6- and 12- month intervals for the radiographic success rate for each caries removal method.

DETAILED DESCRIPTION:
All the lesions in the children's oral cavity indicated for treatment will be treated and sampled for microbiological analysis prior to and following caries removal. On the day of the intervention, the children will be asked to refrain from tooth brushing in the morning, as well as eating and drinking (except water) for at least two hours before the appointment. The patients will be instructed to rinse with a cup of water, then the outer surface of the carious lesion will be washed with a flurry of water to avoid contamination of plaque bacteria. The tooth will then be partially isolated using cotton rolls and saliva ejector.

Two portions of dentin will be collected with sterile excavators from the middle of the cavity to perform the microbiological analysis of each tooth before and then after caries removal procedure. The dentin sample will then be inserted in a sterile test tube containing 1 mL of saline and transported to the microbiology laboratory within 1-2 hours. The bacterial count obtained for a given amount of dentin will be used to estimate the number of colonies present in 1 mg dentin (CFU/mg). In the CMCR group: either Papacarie duo or Brix 3000 gel will be applied on the carious lesion of tooth and left undisturbed for 30-60 seconds, following manufacturer instructions This produces softening of carious dentin, which will be removed with a hand excavator. This step will be repeated 2-3 times until dentin demonstrates slight resistance with no tug-back sensation when tested with an exploratory probe while pressing an explorer into dentin, then the application of the chemo-mechanical agents will be stop The visual test for assessment of complete caries excavation will be based on non-turbid appearance of the CMCR agent used. In the ART group hand excavation will be performed to remove the carious tissue from the cavity by using a sterile sharp hand excavator. The cavity will be determined to be caries-free according to visual and tactile clinical criteria.

No local anesthesia will be administered as it would alter the pain perception of the patient unless necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged 8-10 years old.
2. The presence of at least one deep carious class 1 lesion in the first permanent molar with a score of 5 or 6 according to the International Detection and Assessment System (ICDAS), detected by visual-tactile inspection to assess lesion severity

Exclusion Criteria:

1. Children reporting spontaneous or elicited pain from caries or showing any signs of pulpal infection, swelling or abscess.
2. Pulpal exposure or bleeding during the excavation procedure
3. Children presenting with special health care needs or undergoing medical treatment for chronic or acute diseases affecting salivary flow.
4. Allergy or sensitivity to any of the materials included in the study

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To assess and compare the efficacy of two chemo-mechanical agents Brix 3000 and Papacarie duo in terms of their clinical success in young permanent molars, in comparison with hand excavation approach | one year follow up
  The clinical assessment will be at 3-, 6- and 12-month intervals to evaluate restoration success according to the criteria of atraumatic restorative treatment by Phantumvanit et al. (1996) .Restorations which will receive a score of 0, 1 or 7 will be considered successful while those having a score of 2, 3, 4 or 8 will be considered failures. Those which will receive a score of 5, 6 will be excluded from the analysis.
To assess and compare the efficacy of two chemo-mechanical agents Brix 3000 and Papacarie duo in terms of their radiographic success in young permanent molars, in comparison with hand excavation approach | one year follow up
  The radiographic evaluation will be performed using the radiographic subtraction method

SECONDARY OUTCOMES:
the required time for complete caries removal for each method | immediately after the intervention
  The time needed for complete caries removal will be recorded for each caries removal method.
f patients' subjective pain reactions following each method | immediately after the intervention
  Subjective pain will be assessed after caries removal by means of WongBaker faces scale. It consists of faces with different facial expression for happiness and pain and is scored from 0-5 as 0 is very happy and feels no pain and 5 is very painful
antimicrobial effect of two chemo-mechanical caries removal agents | immediately after the intervention
  Samples from the carious lesion will be collected prior to and following complete caries removal for detection of the change in bacterial count (Streptococci and Lactobacilli counts).

CONTACTS AND LOCATIONS:
Overall Officials: Dalia A Talaat, PHD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol will be availabe
Supporting Information: Study Protocol
Time Frame: June 2023- June 2024
Access Criteria: Researchers interested
URL: http://clinicalTrials.gov

REFERENCES:
- [Derived] Hassanein PH, Samaha AWM, Zakaria AS, Talaat DM. One-year clinical and radiographic evaluation of young permanent molars treated with brix 3000 vs. papacarie duo: a randomized controlled clinical trial. BMC Oral Health. 2025 Sep 23;25(1):1421. doi: 10.1186/s12903-025-06715-7. PMID 40988041